CLINICAL TRIAL: NCT05926349
Title: A Randomized Study of Andexanet Alfa Compared to Usual Care in Patients Receiving a Factor Xa Inhibitor Who Require Urgent Surgery or Procedure (ANNEXA-RS)
Brief Title: A Study of Andexanet Alfa in Patients Requiring Urgent Surgery or Procedure
Acronym: ANNEXA-RS
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Business decision
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D9604C00001
Record Dates: First submitted 2023-06-09; First posted 2023-07-03 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Urgent Surgery
Keywords: Andexanet alfa; Blood Thinners
MeSH Terms: interventions — PRT064445

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Andexanet Alfa Group (Experimental): Patients will receive andexanet alfa as IV bolus followed by an infusion.
  Interventions: Drug: Andexanet alfa
- Usual Care Group (Active Comparator): Patients will receive treatment based on the Investigator's discretion, according to regional, local/institutional guidelines or practices.
  Interventions: Drug: Usual Care

INTERVENTIONS:
Drug: Andexanet alfa — Andexanet is a recombinant version of human FXa
  Other Names: Andexxa®, Ondexxya®
  Arms: Andexanet Alfa Group
Drug: Usual Care — As per the label of the chosen usual care product(s) and/or usual care standards.
  Arms: Usual Care Group

SUMMARY:
The study will aim to find out if the drug andexanet alfa is safe and effective in preventing major bleeding during urgent surgery or invasive procedures. The study will compare the use of andexanet alfa to the usual care given at the study center.

DETAILED DESCRIPTION:
This study will be an open-label, randomised, controlled, prospective, multicenter study. The study will include patients requiring urgent surgery or procedure that needs to be performed within 15 hours of the last dose of blood-thinning drug (direct oral activated Factor X (FXa) inhibitor).

The study will comprise of the following periods:

* Screening, followed by surgery or procedure and study intervention.
* Follow-up period: there will be four follow-up visits over a duration of approximately 30 days.
* Follow-up visit for patients with positive anti-andexanet alfa antibody test: patients with a positive anti-andexanet alfa antibody response at day 30 will have a follow-up anti-andexanet alfa antibody test approximately 120 days post-surgery or procedure.

Patients will be randomised in the ratio of 1:1 to receive either andexanet alfa or usual care.

ELIGIBILITY:
Inclusion Criteria:

* The patient requires, in the opinion of the Investigator, urgent surgery or procedure and requires reversal of direct oral FXa inhibition.
* The patient requires urgent surgery or procedure within 12 hours of informed consent.
* The patient requires urgent surgery or procedure that is expected to be associated with a high risk of bleeding or bleeding to occur into a critical organ.
* The patient has taken an oral FXa inhibitor (such as apixaban, rivaroxaban, or edoxaban) within 15 hours or more, prior to start of surgery or procedure.
* Female patients of childbearing potential must have a negative pregnancy test at Screening.
* Willingness to use highly effective methods of contraception (for male and female patients who are fertile).

Exclusion Criteria:

* The patient requires surgeries or procedures that have a very low chance of causing significant, uncontrollable bleeding, such as small skin procedures, cataract surgery, and minor dental procedures.
* The patient has acute life-threatening bleeding at the time of Screening.
* The patient will undergo a surgery or procedure which will require the use of heparin.
* Patient who is not expected to live for more than three months due to other health problems or has specifically requested not to be resuscitated if their heart stops beating.
* Prior to screening, the patient had either experienced low platelet count due to heparin use with or without blood clots or had a genetic condition that affects blood clotting.
* Patient has acute decompensated heart failure, cardiogenic shock, sepsis, or septic shock at the time of Screening.
* Patient has history of heparin-induced thrombocytopenia (with or without thrombosis) or inherited coagulopathy (eg, anti-thrombin III deficiency, anti-phospholipid antibody syndrome, protein C/S deficiency, Factor V Leiden) at the time of Screening.
* Previously diagnosed with a bleeding disorder (eg, platelet function disorder, hemophilia, Von Willebrand disease, or coagulation factor deficiency).
* Prior known hypersensitivity to andexanet alfa.
* Use of andexanet alfa 30 days prior to Screening.
* Patient diagnosed with dementia.
* Any prohibited medication as determined in the study.

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-08-02 (Estimated); Primary Completion 2027-01-05 (Estimated); Study Completion 2027-09-07 (Estimated)

PRIMARY OUTCOMES:
Number of patients achieving effective intraoperative hemostasis | From start to the end of surgery or procedure on Day 0
  Intraoperative hemostasis will be assessed according to the categories as per 4-point hemostasis scale: Excellent - Normal hemostasis, Good - Mildly abnormal hemostasis (eg. slight oozing from surgical wounds), Moderate - Moderate abnormality in intraprocedural hemostasis (eg. controllable bleeding), Poor - Severe hemostatic abnormality (eg. severe refractory hemorrhage). Hemostasis will be considered to be effective if the intraoperative hemostasis category is 'excellent' or 'good', and ineffective if the intraoperative hemostasis category is 'moderate' or 'poor'.

SECONDARY OUTCOMES:
Change from Baseline in anti-FXa activity measured through blood samples | Baseline to start of surgery or procedure
  The ability of andexanet alfa to rapidly reverse the anticoagulation effect of FXa inhibitors by reduction of anti-FXa activity when compared to usual care.
Change from Baseline in anti-FXa activity measured through blood samples | Baseline to two hours post start of surgery or procedure
  The ability of andexanet alfa to sustainably reverse the anticoagulation effect of FXa inhibitors by reduction of anti-FXa activity when compared to usual care at two hours post start of surgery or procedure will be assessed.

OTHER OUTCOMES:
Number of patients with adverse events | Screening (Day -1 to Day 0) until follow-up visit (Day 30 or Day 120)
  Safety and tolerability will be evaluated in terms of adverse events and serious adverse events.

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All requests will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com /ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please refer to our disclosure commitment at:
  https://astrazenecagrouptrials.pharmacm.com /ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patientlevel data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at:
  https://astrazenecagrouptrials.pharmacm.com /ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home